CLINICAL TRIAL: NCT01522040
Title: A Pilot Study of Magnesium Infusions (Drips) for Moderate-to-Severe Pediatric Asthma Exacerbations
Brief Title: Pilot Study of Magnesium Infusions in Pediatric Asthma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Keith Cross, Assistant Professor of Pediatrics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11.0641
Record Dates: First submitted 2012-01-24; First posted 2012-01-31 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; Magnesium; Adrenergic Receptor
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium (Active Comparator): Half the enrolled subjects will be randomized to receive active drug, a magnesium infusion.
  Interventions: Drug: Magnesium Sulfate
- Control (Placebo Comparator): Half the subjects will be randomized to receive a drip that does not have active drug (magnesium sulfate).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — Continuous magnesium drip, titrated to effect until patient's symptoms improve
  Arms: Magnesium
Drug: Placebo — Simple saline drip, without active drug
  Arms: Control

SUMMARY:
This is a prospective randomized pilot study that seeks to address the research question: In children with moderate-to-severe asthma, do intravenous magnesium infusions added to standard Pediatric intensive care unit (PICU)-level asthma care significantly decrease time from patient presentation until PICU discharge?

DETAILED DESCRIPTION:
This study will be a double-blind, prospective randomized pilot study. Subjects will be randomized on a 1:1 basis to receive routine asthma care with or without a magnesium drip.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 years 0 days up to 20 years 364 days
* Clinical diagnosis of asthma including both of the following:

  * Attending physician's primary working diagnosis is status asthmaticus
  * Results of a modified International Study of Asthma and Allergies in Children (ISAAC) diagnostic questionnaire consistent with an asthma diagnosis
* Planned PICU admission for moderate-to-severe asthma exacerbation persisting despite standard first-tier therapy (systemic corticosteroids and at least a one-hour treatment with nebulized albuterol/ipratroprium or equivalent) as evidenced by an asthma score of 7 or greater
* IV access or equivalent
* Ability to understand and give informed consent/assent in English

Exclusion Criteria:

* Prior enrollment in this study
* Prior adverse reactions to magnesium
* Use of systemic corticosteroids or magnesium in preceding 2 weeks, or administered at a transferring facility more than 3 hours prior to enrollment
* Admission for inpatient asthma care in preceding 2 weeks
* Hemodynamic instability, impending respiratory failure or intubation
* Inability in children age 7 years or older to give assent due to a developmental delay or altered mental status
* Significant renal or cardiac disease
* Sickle cell anemia
* Significant, active non-asthma pulmonary disease

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Time to discharge | Duration of hospital stay, typically 3-5 days
  The primary outcome for this study is elapsed time from emergency department (ED) presentation to readiness for PICU discharge.

SECONDARY OUTCOMES:
Beta receptor haplotype | Once on enrollment
  The subject's genetic haplotype for beta adrenergic receptor. It will be determined by blood test during their admission in the hospital and enrollment on the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cross, MD, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States